CLINICAL TRIAL: NCT04498247
Title: A Phase 1/Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Trial to Evaluate the Safety, Tolerability and Immunogenicity of V591 (COVID-19 Vaccine) in Healthy Younger and Older Participants
Brief Title: A Study to Assess Safety, Tolerability, and Immunogenicity of V591 (COVID-19 Vaccine) in Healthy Participants (V591-001)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on an interim assessment of immunogenicity
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: V591-001; 2020-003493-46 (EudraCT Number); V591-001 (Other: Merck)
Record Dates: First submitted 2020-08-03; First posted 2020-08-04 (Actual); Results first posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Panel A (Experimental): Participants in this 18 to 55 year old sentinel cohort will receive 2 doses (Day 1 and Day 57) of 1x10^5 50% tissue culture infectious dose (TCID50) V591 or placebo
  Interventions: Biological: V591; Other: Placebo
- Panel B (Experimental): Participants in this 18 to 55 year old sentinel cohort will receive 2 doses (Days 1 and 57) of 1x10^6 TCID50 V591 or placebo
  Interventions: Biological: V591; Other: Placebo
- Panels C, G (Experimental): Participants in this 18 to 55 year old cohort (Panel C) or >55 year old cohort (Panel G) will receive 1 dose of 1x10^5 TCID50 V591 or placebo.
  Interventions: Biological: V591; Other: Placebo
- Panels D, H (Experimental): Participants in this 18 to 55 year old cohort (Panel D) or >55 year old cohort (Panel H) will receive 1 dose of 1x10^6 TCID50 V591 or placebo.
  Interventions: Biological: V591; Other: Placebo
- Panel E (Experimental): Participants in this 18 to 55 year old cohort will receive 1 dose of 1x10^7 V591 or placebo.
  Interventions: Biological: V591; Other: Placebo
- Panel F (Experimental): Participants in this 18 to 55 year old cohort will receive 2 doses (Days 1 and 169) of V591 or placebo. Day 1 will be 1x10^4 TCID50 V591 or placebo and Day 169 will be 1x10^5 TCID50 V591 or placebo.
  Interventions: Biological: V591; Other: Placebo
- Panel I (Experimental): Participants in this >55 year old cohort will receive 2 doses (Days 1 and 57) of 1x10^5 TCID50 V591 or placebo
  Interventions: Biological: V591; Other: Placebo
- Panel J (Experimental): Participants in this >55 year old cohort will receive 2 doses (Days 1 and 57) of 1x10^6 TCID50 V591 or placebo
  Interventions: Biological: V591; Other: Placebo
- Panel K (Experimental): Participants in this >55 year old cohort will receive 2 doses (Days 1 and 169) of 1x10^5 TCID50 V591 or placebo
  Interventions: Biological: V591; Other: Placebo
- Panel L (Experimental): Participants in this >55 year old cohort will receive 2 doses (Days 1 and 169) of 1x10^6 TCID50 V591 or placebo
  Interventions: Biological: V591; Other: Placebo

INTERVENTIONS:
Biological: V591 — 1 or 2 ascending doses of V591 will be administered via intramuscular (IM) injection.
Other: Placebo — Placebo (0.9% sodium chloride) administered via IM injection.

SUMMARY:
The primary objective of this early Phase 1/2 study is to identify the V591 dose that achieves the target immune response in humans based on preclinical or early clinical data.

DETAILED DESCRIPTION:
This study was terminated and modifications to the dosing regimens and clinical/laboratory procedures were implemented for trial discontinuation according to Protocol Amendment 04. Per protocol, certain panels were never enrolled and/or the second dose of study intervention was not administered.

ELIGIBILITY:
Inclusion Criteria:

* Is in overall good health based on medical history, physical examination, electrocardiogram (ECG) and vital sign (VS) measurements performed prior to randomization.
* Is in overall good health based on laboratory safety tests obtained at the screening visit.
* Has a body mass index (BMI) <30 kg/m2 inclusive. On this basis a rounded BMI of 29.9 is acceptable to satisfy the inclusion criteria. BMI = weight (kg)/height (m)2.
* Has been practicing social distancing for at least two weeks prior to planned Day 1 vaccination and has no close contacts with known active severe acute respiratory syndrome coronavirus (SARS-CoV)-2 infection in that time period.
* Sentinel trial participants ONLY (Panel A, Panel B, and the first 5 participants of Panel E): Seronegative for SARS-COV-2.
* Is male or female, from 18 years to 55 years of age (inclusive) (Parts 1 and 2A) or >55 years of age (Part 2B), at the time of providing documented informed consent.
* Male participants are eligible to participate if they agree to refrain from donating sperm during the intervention period and for at least 6 months after the last dose of study intervention, be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent OR agree to use contraception unless confirmed to be azoospermic .
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, is not a woman of childbearing potential (WOCBP) or Is a WOCBP and using an acceptable contraceptive method or be abstinent from heterosexual intercourse as their preferred and usual lifestyle.
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) before the first dose of study intervention. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* Refrain from donating oocyte during the intervention period and for at least 6 months after the last dose of study intervention.
* The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* The participant (or legally acceptable representative) has provided documented informed consent/assent for the study, including for future biomedical research.
* Is willing to comply with the study restrictions, including social distancing between screening and randomization.
* Is willing to abstain from donating whole blood or blood derivatives, tissue or organ all along the study.
* Agrees to provide study personnel with a primary telephone number as well as an alternate means of contact, if available (such as an alternate telephone number or email) for follow-up purposes.
* Can read, understand, and complete the Vaccination Report Card.

Exclusion Criteria

* Is currently actively infected with SARS-CoV-2 (confirmed by polymerase chain reaction;[PCR]).
* Has prior medical history of confirmed SARS-CoV-2 infection or known exposure to an individual with confirmed coronavirus disease 2019 (COVID-19) disease or SARS CoV-2 infection within the past 2 weeks. With the exception of the sentinel participants (Panel A, Panel B, and the first 5 participants of Panel E), study participants will not be screened for enrollment by SARS-CoV-2 serology, allowing those who may have had a prior asymptomatic SARS-CoV-2 infection to be enrolled.
* Has a history of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as urticaria, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of known or suspected allergic reaction likely to be exacerbated by any component of the COVID-19 vaccine.
* Is currently (or highly suspected to be) immunocompromised, including anticipating the need for systemic immunosuppressive treatment within the next 6 months or 12 months for 2-dose Day 1, Day 169 panels or has been diagnosed or highly suspected as having a congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune condition that could impact the immune response or the safety of the study vaccine.
* Has clinically significant thrombocytopenia or other coagulation disorder contraindicating intramuscular vaccination or repeated venipuncture.
* Has history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might expose the participant to risk by participating in the study, confound the results of the study or interfere with the participant's participation for the full duration of the study.
* Has a history or presence of clinically significant pulmonary disorders (e.g. chronic obstructive pulmonary disease [COPD], etc.), or asthma.
* Has a history of confirmed SARS-CoV-1 or Middle Eastern respiratory syndrome (MERS)
* Has a history of or current clinically significant medical condition that puts or may put a participant at increased risk for severe SARS-CoV-2 disease, such as conditions associated with increased risk of severe illness from COVID-19, cancer, chronic kidney disease, COPD, immunocompromised state (weakened immune system) from solid organ transplant, obesity (BMI of 30 or higher), serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies, sickle cell disease, Type 2 diabetes mellitus, asthma, cerebrovascular disease, cystic fibrosis, hypertension or high blood pressure, an immunocompromised state (weakened immune system), neurologic conditions, such as dementia, liver disease, pregnancy, pulmonary fibrosis (having damaged or scarred lung tissues), smoking, thalassemia (a type of blood disorder), or Type 1 diabetes mellitus.
* Part 2B ONLY: Older adult participants having mild, well controlled hypertension as is widely characteristic of aging are allowed if their medication regimens have not substantively changed for the past 6 months, hypertension has not led to hospitalization or currently increased rate of clinic visits over the past year, and hypertension has not been confirmed as putting subjects at increased risk of severe illness from COVID-19 by the CDC (https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/groups-at-higher-risk.html).
* Is mentally or legally incapacitated, has significant emotional problems at the time of pre-study (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years.
* Has a history of any clinically significant major neurological disorders or seizures (including Guillain-Barré syndrome), with the exception of febrile seizures during childhood.
* Has a history of cancer (malignancy)
* Has a known or suspected history of significant multiple and/or severe allergies (e.g., food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e., systemic allergic reaction) to prescription or non-prescription drugs or food.
* Is positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV)-1 or 2 antibodies. Individuals with antibodies to hepatitis C may be enrolled if hepatitis C viral load is undetectable and there is no evidence of or history of liver disease.
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pre-study (screening) visit.
* Has received immunosuppressive drugs (like e.g. systemic corticosteroids, excluding topical preparations and inhalers) within 3 months prior to the first vaccination or 6 months for chemotherapies.
* *Has received vaccination within 4 weeks prior to first vaccination or is planning to receive a licensed vaccine 4 weeks before or after each study vaccination (e.g.

Inactivated influenza vaccine).

* *Has received measles-containing vaccine within 3 months prior to the first vaccination.
* Has received a blood transfusion or blood products, including immunoglobulin, starting from 3 months before the first study vaccination or is scheduled to receive a blood transfusion or blood product through study completion. Autologous blood transfusions are not considered an exclusion criterion.
* Is unable to meet the concomitant medication restrictions
* Is using antiviral medications or any investigational agents for prophylaxis of SARSCoV-2 within 4 weeks prior to the first vaccination.
* Has ever participated in an investigational study of a SARS-CoV-2 vaccine, or an antiviral or other biologic product intended for the treatment of COVID-19.
* Is currently participating in any study of a vaccine or investigational medicinal product (IMP) or has recently completed participation in another study of a vaccine or IMP and received a vaccine within 3 months prior to screening or an IMP within 4 weeks (or 5 half-lives of the IMP, whichever is longer) prior to the pre-study (screening) visit. The window will be derived from the date of the last study intervention (e.g., receiving a vaccine or IMP) in the previous study to the date of the pre-study (screening) visit for this study. In addition, a participant cannot participate in another investigational trial up to the post-trial visit of this study (approximately 12 months after the last study vaccination).
* Has glycated hemoglobin (A1C) ≥ 6.5% at screening.
* Has a history of alcohol, cocaine, or opioid abuse during the previous 3 years.
* Participants who currently smoke or used nicotine or nicotine-containing products (e.g. nicotine patch) within last 3 months. Former smokers that have less than a 10 pack-year history of smoking and have not smoked in the last 12 months are eligible to be enrolled.
* Has a tattoo, scar or other physical finding at the area of the vaccination site that would interfere with intramuscular injection or a local tolerability assessment.
* Presents any concern by the investigator regarding safe participation in the study or for any other reason the investigator considers the participant inappropriate for participation in the study.
* Lives in a nursing home or long-term care facility.
* Is currently working in occupations with high risk of exposure to SARS-CoV-2 (e.g., health care worker with direct patient contact, emergency response personnel), or, at the investigator's discretion to be at increased risk to acquire SARS-CoV-2 for any other reason.
* Individuals who are living and/or working with severely immunocompromised people, pregnant women, lactating women, children under 12 months old, or any other individual that, in the judgment of the investigator, might be at increased risk.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigatively involved with this study.

  * if the participant meets these exclusion criteria, the Day 1 Visit may be rescheduled for a time when these criteria are not met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (9):
- United States (4):
  - Research Centers of America, LLC ( Site 0014), Hollywood, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0013), Wichita, Kansas
  - Central Kentucky Research Associates, Inc. ( Site 0011), Lexington, Kentucky
  - The Center for Pharmaceutical Research PC ( Site 0012), Kansas City, Missouri
- Austria (2):
  - SCRI-CCCIT GesmbH ( Site 0006), Salzburg
  - Medizinische Universitaet Wien ( Site 0007), Vienna
- Belgium (3):
  - Universitair Ziekenhuis Gent ( Site 0003), Ghent, Oost-Vlaanderen
  - SGS Life Science Services ( Site 0001), Antwerp
  - ATC - Clinical Pharmacology Unit ( Site 0002), Liège

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Vanhoutte F, Liu W, Wiedmann RT, Haspeslagh L, Cao X, Boundy K, Aliprantis A, Davila M, Hartzel J, Li J, McGuire M, Ramsauer K, Tomberger Y, Tschismarov R, Brown DD, Xu W, Sachs JR, Russell K, Stoch SA, Lai E. Safety and immunogenicity of the measles vector-based SARS-CoV-2 vaccine candidate, V591, in adults: results from a phase 1/2 randomised, double-blind, placebo-controlled, dose-ranging trial. EBioMedicine. 2022 Jan;75:103811. doi: 10.1016/j.ebiom.2021.103811. Epub 2022 Jan 15. PMID 35042081

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults with no prior history of confirmed Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection, or known exposure to an individual with confirmed Coronavirus Disease 2019 (COVID-19) or SARS-CoV-2 infection were enrolled in this study.
Groups:
- V591 1×10^4 TCID50-1 Dose: Participants received one dose of V591 1x10^4 tissue culture infectious dose (TCID50) on Day 1
- V591 1×10^5 TCID50-1 Dose: Participants received one dose of V591 1×10^5 TCID50 on Day 1.
- V591 1x10^5 TCID50- 2 Dose: Participants received one dose of V591 1×10^5 TCID50 on Day 1 and a second V591 1×10^5 TCID50 dose on Day 57.
- V591 1×10^6 TCID50-1 Dose: Participants received one dose of V591 1×10^6 TCID50 on Day 1
- V591 1×10^6 TCID50-2 Dose: Participants received one dose of V591 1×10^6 TCID50 on Day 1 and a second V591 1×10^6 TCID50 dose on Day 57.
- V591 1×10^7 TCID50: Participants received one dose of V591 1×10^7 TCID50 on Day 1
- Placebo- 1 Dose: Participants received one dose of placebo on Day 1
- Placebo- 2 Dose: Participants received one dose of placebo on Day 1 and a second dose of placebo on Day 57.
Period: Overall Study
Arm/Group | V591 1×10^4 TCID50-1 Dose | V591 1×10^5 TCID50-1 Dose | V591 1x10^5 TCID50- 2 Dose | V591 1×10^6 TCID50-1 Dose | V591 1×10^6 TCID50-2 Dose | V591 1×10^7 TCID50 | Placebo- 1 Dose | Placebo- 2 Dose
Started | 21 | 80 | 4 | 81 | 4 | 20 | 51 | 2
Vaccination 1 | 20 | 80 | 4 | 81 | 4 | 20 | 51 | 2
Vaccination 2 | 0 | 0 | 4 | 0 | 4 | 0 | 0 | 2
Completed | 20 | 68 | 4 | 70 | 4 | 20 | 43 | 2
Not Completed | 1 | 12 | 0 | 11 | 0 | 0 | 8 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Mistakenly Randomized; Not Treated | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 8 | 0 | 7 | 0 | 0 | 1 | 0
Not completed — Received a non-study COVID-19 vaccine. | 0 | 4 | 0 | 3 | 0 | 0 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- V591 1×10^4 TCID50-1 Dose: Participants received one dose of V591 1x10^4 TCID50 on Day 1
- V591 1×10^5 TCID50- 1 Dose: Participants received one dose of V591 1×10^5 TCID50 on Day 1.
- Placebo - 1 Dose: Participants received one dose of placebo on Day 1.
- Total: Total of all reporting groups
Arm/Group | V591 1×10^4 TCID50-1 Dose | V591 1×10^5 TCID50- 1 Dose | V591 1x10^5 TCID50- 2 Dose | V591 1×10^6 TCID50-1 Dose | V591 1×10^6 TCID50-2 Dose | V591 1×10^7 TCID50 | Placebo - 1 Dose | Placebo- 2 Dose | Total
Number analyzed (Participants) | 21 | 80 | 4 | 81 | 4 | 20 | 51 | 2 | 263
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.7 (10.4) | 59.7 (14.8) | 45.0 (6.6) | 58.4 (15.2) | 40.3 (13.2) | 26.6 (6.8) | 56.2 (17.9) | 34.5 (0.7) | 53.8 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 46 | 3 | 43 | 4 | 14 | 27 | 2 | 148
  Male | 12 | 34 | 1 | 38 | 0 | 6 | 24 | 0 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 20 | 0 | 12 | 1 | 0 | 3 | 0 | 37
  Not Hispanic or Latino | 20 | 60 | 4 | 69 | 3 | 20 | 48 | 2 | 226
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 5
  White | 19 | 77 | 4 | 78 | 4 | 20 | 50 | 2 | 254
  More than one race | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Solicited Injection Site Adverse Event (AE) After Any Study Intervention
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Injection site AEs of pain/tenderness, swelling, and redness/erythema were assessed.
Time Frame: Up to 5 days after any study intervention
Population: All randomized participants who received at least one dose of study intervention and received the dose relevant to the data collection time point. Participants were pooled by dose of study intervention administered due to the study's termination prior to most participants receiving their planned second dose.
Measure: Number; unit: Percentage of participants
Groups:
- V591 1×10^4 TCID50: Participants received one dose of V591 1x10^4 TCID50 on Day 1
- V591 1×10^5 TCID50: All participants received one dose of V591 1×10^5 TCID50 on Day 1; Some participants received a second V591 1×10^5 TCID50 dose on Day 57.
- V591 1×10^6 TCID50: All participants received one dose of V591 1×10^6 TCID50 on Day 1; Some participants received a second V591 1×10^6 TCID50 dose on Day 57.
- Placebo: Participants received one dose of placebo on Day 1; Some participants received a second dose of placebo on Day 57.
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
Percentage of participants
  Following Vaccination 1 | 25.0 | 6.0 | 15.3 | 55.0 | 7.5
  Following Vaccination 2: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Following Vaccination 2 |  | 0.0 | 25.0 |  | 0.0

2. Primary Outcome: Percentage of Participants With at Least One Solicited Systemic AE After Any Study Intervention
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Systemic AEs of fever, muscle pain, joint pain, headache, fatigue, rash, or nausea were assessed.
Time Frame: Up to 14 days after any study intervention
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
Percentage of participants
  Following Vaccination 1 | 50.0 | 45.2 | 37.6 | 65.0 | 56.6
  Following Vaccination 2: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Following Vaccination 2 |  | 25.0 | 75.0 |  | 50.0

3. Primary Outcome: Percentage of Participants With at Least One Unsolicited Adverse Event After Any Study Intervention
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. All unsolicited AEs were assessed.
Time Frame: Up to 28 days after any study intervention
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
Percentage of participants
  Following Vaccination 1 | 55.0 | 34.5 | 32.9 | 70.0 | 37.7
  Following Vaccination 2: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Following Vaccination 2 |  | 0.0 | 25.0 |  | 0.0

4. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event
Description: An SAE is defined as any untoward medical occurrence that at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Up to 56 days after vaccination 1 and up to 122 days after vaccination 2 (up to 178 days)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
Percentage of Participants
  Following Vaccination 1 | 0.0 | 0.0 | 2.4 | 0.0 | 1.9
  Following Vaccination 2: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Following Vaccination 2 |  | 0.0 | 0.0 |  | 0.0

5. Primary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an Adverse Event
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 57 days
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
Percentage of Participants
  Following Vaccination 1 | 5.0 | 6.0 | 4.7 | 0 | 5.7
  Following Vaccination 2: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Following Vaccination 2 |  | 0.0 | 0.0 |  | 0.0

6. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended Adverse Event (MAAE)
Description: A MAAE is defined as an adverse event in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency room visit, office visit, or an urgent care visit with any medical personnel for any reason.
Time Frame: Up to 56 days after vaccination 1 and up to 122 days after vaccination 2 (up to 178 days)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
Percentage of Participants
  Following Vaccination 1 | 30.0 | 10.7 | 11.8 | 40.0 | 9.4
  Following Vaccination 2: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Following Vaccination 2 |  | 0.0 | 0.0 |  | 0.0

7. Secondary Outcome: Geometric Mean Titers for Serum Neutralizing Antibodies (nAb) as Measured by Pseudo-virus Neutralization Assay (PNA)
Description: Serum samples were collected and the titers of serum neutralization antibodies were assessed using PNA. Geometric mean titers were calculated using a constrained longitudinal data analysis (cLDA) method where the response vector consisted of the log transformed pre-vaccination and post-vaccination antibody titers. The point estimates were calculated by exponentiating the estimates of the mean of the natural log values; and the within-group 95% confidence intervals (CIs) were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Days 1, 15, 29, 57, 71, and 85
Population: All randomized participants without deviations from the protocol that may substantially affect the results of the immunogenicity endpoint, and who had available data at the indicated time point. Participants were pooled by dose of study intervention administered due to the study's termination prior to most participants receiving their planned second dose. Data were not collected for planned timepoints on days 115, 211, 365, 422, and 534 due to early termination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
Titer
  Day 1: number analyzed (Participants) | 20 | 84 | 84 | 20 | 51
  Day 1 | 5.0 [5.0 to 5.0] | 6.3 [5.1 to 7.8] | 5.9 [5.0 to 6.9] | 9.1 [5.0 to 16.7] | 5.0 [5.0 to 5.0]
  Day 15: number analyzed (Participants) | 19 | 84 | 78 | 20 | 47
  Day 15 | 5.8 [4.2 to 8.1] | 6.7 [5.3 to 8.5] | 7.9 [6.1 to 10.4] | 53.1 [17.2 to 164.6] | 5.3 [4.7 to 6.1]
  Day 29: number analyzed (Participants) | 20 | 79 | 81 | 20 | 50
  Day 29 | 5.0 [5.0 to 5.0] | 8.3 [6.0 to 11.3] | 8.3 [6.3 to 11.0] | 31.2 [11.2 to 86.7] | 6.3 [4.8 to 8.1]
  Day 57: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 57 |  | 13.7 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 5.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 5.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.
  Day 71: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 71 |  | 25.7 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 45.2 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 5.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.
  Day 85: number analyzed (Participants) | 0 | 4 | 3 | 0 | 2
  Day 85 |  | 24.6 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 54.2 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 5.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.

8. Secondary Outcome: Geometric Mean Concentration of Total Anti-Spike Immunoglobulin G (IgG) Antibodies as Measured by Enzyme-Linked Immunosorbent Assay (ELISA)
Description: Serum samples were collected and the concentrations of total anti-spike IgG antibodies were assessed using ELISA. Geometric mean concentrations were calculated using a cLDA method where the response vector consisted of the log transformed pre-vaccination and post-vaccination antibody titers. The point estimates were calculated by exponentiating the estimates of the mean of the natural log values; and the within-group 95% confidence intervals (CIs) were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Days 1, 15, 29, 57, 71, and 85
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA unit/mL
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
ELISA unit/mL
  Day 1: number analyzed (Participants) | 20 | 84 | 82 | 20 | 51
  Day 1 | 25.2 [25.2 to 25.2] | 33.9 [26.1 to 44.0] | 36.3 [28.2 to 46.9] | 46.3 [24.7 to 86.8] | 26.1 [24.8 to 27.5]
  Day 15: number analyzed (Participants) | 19 | 84 | 76 | 20 | 47
  Day 15 | 26.2 [24.1 to 28.5] | 35.7 [27.2 to 46.7] | 41.6 [30.0 to 57.6] | 239.2 [78.8 to 725.9] | 26.4 [24.7 to 28.2]
  Day 29: number analyzed (Participants) | 20 | 79 | 79 | 20 | 50
  Day 29 | 28.6 [23.7 to 34.6] | 44.0 [31.6 to 61.3] | 52.6 [36.6 to 75.6] | 294.8 [110.3 to 788.2] | 31.5 [25.3 to 39.3]
  Day 57: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 57 |  | 97.7 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 25.2 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 25.2 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.
  Day 71: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 71 |  | 184.7 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 336.1 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 25.2 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.
  Day 85: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 85 |  | 180.8 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 260.6 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 25.2 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.

9. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Serum nAb as Measured by PNA
Description: Serum samples were collected and the titers of serum neutralization antibodies were assessed using PNA. Geometric mean titers were calculated using a cLDA method where the response vector consisted of the log transformed pre-vaccination and post-vaccination antibody titers. GMFR is defined as the geometric mean of the ratio of concentration at specified timepoints after vaccination divided by concentration at baseline (Day 1).
Time Frame: Days 1, 15, 29, 57, 71, and 85
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
Ratio
  Day 15: number analyzed (Participants) | 19 | 84 | 78 | 20 | 47
  Day 15 | 1.1 [0.9 to 1.4] | 1.0 [1.0 to 1.1] | 1.2 [1.1 to 1.5] | 4.1 [2.0 to 8.3] | 1.1 [0.9 to 1.2]
  Day 29: number analyzed (Participants) | 20 | 79 | 81 | 20 | 50
  Day 29 | 1.0 [1.0 to 1.0] | 1.2 [1.0 to 1.5] | 1.3 [1.1 to 1.6] | 2.6 [1.2 to 5.5] | 1.2 [1.0 to 1.5]
  Day 57: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 57 |  | 2.3 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 1.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 1.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.
  Day 71: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 71 |  | 3.6 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 4.5 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 1.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.
  Day 85: number analyzed (Participants) | 0 | 4 | 3 | 0 | 2
  Day 85 |  | 3.5 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 5.4 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 1.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.

10. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Total Anti-Spike IgG Antibodies as Measured by ELISA
Description: Serum samples were collected and the total anti-spike IgG antibodies assessed using ELISA. Geometric mean concentrations were calculated using a cLDA method where the response vector consisted of the log transformed pre-vaccination and post-vaccination antibody titers. GMFR is defined as the geometric mean of the ratio of concentration at specified timepoints after vaccination divided by concentration at baseline (Day 1).
Time Frame: Days 1, 15, 29, 57, 71, and 85
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V591 1×10^4 TCID50 | V591 1×10^5 TCID50 | V591 1×10^6 TCID50 | V591 1×10^7 TCID50 | Placebo
Number analyzed (Participants) | 20 | 84 | 85 | 20 | 53
Ratio
  Day 15: number analyzed (Participants) | 19 | 84 | 76 | 20 | 47
  Day 15 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.3] | 3.5 [1.8 to 6.9] | 1.0 [0.9 to 1.0]
  Day 29: number analyzed (Participants) | 20 | 79 | 79 | 20 | 50
  Day 29 | 1.1 [1.0 to 1.2] | 1.2 [1.0 to 1.4] | 1.3 [1.1 to 1.6] | 3.9 [1.8 to 8.6] | 1.2 [1.0 to 1.4]
  Day 57: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 57 |  | 3.3 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 1.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 1.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.
  Day 71: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 71 |  | 5.2 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 6.7 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 1.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.
  Day 85: number analyzed (Participants) | 0 | 4 | 4 | 0 | 2
  Day 85 |  | 5.1 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. | 5.2 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants. |  | 1.0 [NA to NA] — The 95% confidence interval is not provided when n is less than 5 participants.

ADVERSE EVENTS:
Time Frame: Serious adverse events and all cause mortality were collected throughout the duration of the study (up to day 178). Non-serious adverse events were assessed up to day 146.
Description: The analysis population for all cause mortality consists of all randomized participants. The analysis populations for serious and non-serious adverse events include all randomized participants who received at least one dose of study intervention. Adverse events were reported separately by occurrence after the first dose of study intervention or second dose of study intervention.
Groups:
- V591 1x10⁴ TCID₅₀-Post Vaccination (Vacc) 1: Participants received one dose of 1x10^4 TCID50 V591 on Day 1
- V591 1x10⁵ TCID₅₀-Post Vacc 1: All participants received one dose of V591 1×10^5 TCID50 on Day 1; Some participants received a second V591 1×10^5 TCID50 dose on Day 57.
- V591 1x10⁶ TCID₅₀-Post Vacc 1: All participants received one dose of V591 1×10^6 TCID50 on Day 1; Some participants received a second V591 1×10^6 TCID50 dose on Day 57.
- V591 1x10⁷ TCID₅₀-Post Vacc 1: Participants received one dose of V591 1×10^7 TCID50 on Day 1
- Placebo-Post Vacc 1: Participants received one dose of placebo on Day 1; Some participants received a second dose of placebo on Day 57.
- V591 1x10⁵ TCID₅₀-Post Vacc 2: All participants received 2 doses of V591; one dose of V591 1×10^5 TCID50 on Day 1 and a second dose of V591 1×10^5 TCID50 on Day 57.
- V591 1x10⁶ TCID₅₀-Post Vacc 2: All participants received 2 doses of V591; one dose of V591 1×10^6 TCID50 on Day 1 and a second dose of V591 1×10^6 TCID50 on Day 57.
- Placebo-Post Vacc 2: All participants received 2 doses of placebo; one dose of placebo on Day 1 and a second dose of placebo on Day 57.
Arm/Group | V591 1x10⁴ TCID₅₀-Post Vaccination (Vacc) 1 | V591 1x10⁵ TCID₅₀-Post Vacc 1 | V591 1x10⁶ TCID₅₀-Post Vacc 1 | V591 1x10⁷ TCID₅₀-Post Vacc 1 | Placebo-Post Vacc 1 | V591 1x10⁵ TCID₅₀-Post Vacc 2 | V591 1x10⁶ TCID₅₀-Post Vacc 2 | Placebo-Post Vacc 2
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/84 | 0/85 | 0/20 | 0/53 | 0/4 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/84 | 2/85 | 0/20 | 1/53 | 0/4 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 15/20 | 47/84 | 41/85 | 20/20 | 35/53 | 1/4 | 3/4 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V591 1x10⁴ TCID₅₀-Post Vaccination (Vacc) 1 (N=20) | V591 1x10⁵ TCID₅₀-Post Vacc 1 (N=84) | V591 1x10⁶ TCID₅₀-Post Vacc 1 (N=85) | V591 1x10⁷ TCID₅₀-Post Vacc 1 (N=20) | Placebo-Post Vacc 1 (N=53) | V591 1x10⁵ TCID₅₀-Post Vacc 2 (N=4) | V591 1x10⁶ TCID₅₀-Post Vacc 2 (N=4) | Placebo-Post Vacc 2 (N=2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V591 1x10⁴ TCID₅₀-Post Vaccination (Vacc) 1 (N=20) | V591 1x10⁵ TCID₅₀-Post Vacc 1 (N=84) | V591 1x10⁶ TCID₅₀-Post Vacc 1 (N=85) | V591 1x10⁷ TCID₅₀-Post Vacc 1 (N=20) | Placebo-Post Vacc 1 (N=53) | V591 1x10⁵ TCID₅₀-Post Vacc 2 (N=4) | V591 1x10⁶ TCID₅₀-Post Vacc 2 (N=4) | Placebo-Post Vacc 2 (N=2)
Nausea (Gastrointestinal disorders) | 3 (6) | 7 (9) | 2 (2) | 4 (4) | 7 (8) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (14) | 22 (30) | 19 (25) | 8 (13) | 20 (26) | 1 (1) | 2 (2) | 0 (0)
Injection site movement impairment (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 5 (5) | 6 (6) | 13 (14) | 11 (11) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 9 (9) | 8 (8) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 8 (10) | 7 (8) | 1 (1) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 14 (15) | 14 (15) | 3 (3) | 10 (14) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 24 (34) | 20 (31) | 9 (16) | 19 (22) | 0 (0) | 2 (3) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated based on an interim assessment of immunogenicity indicating that V591 was not predicted to provide adequate protection against disease caused by SARS-CoV-2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04498247/Prot_SAP_000.pdf